CLINICAL TRIAL: NCT05247775
Title: Urethral Functional Profile Length Before Radical Prostatectomy as an Early Postoperative Continence Predictor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Mirko Bakula, Urology specialist, Clinical Hospital Centre Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25062009
Record Dates: First submitted 2022-02-04; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; Radical Prostatectomy; Urethral Pressure Profile; ICIQ-UI SF; Pads
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with prostate cancer (Experimental): We performed urethral pressure profilometry prior to open retropubic radical prostatectomy (ORRP). Patients were interviewed about the urinary incontinence by the usage of pads and International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) prior to ORRP and at 2, 8, 16 and 24 weeks after ORRP.
  Interventions: Procedure: Profilometry

INTERVENTIONS:
Procedure: Profilometry — Profilometry was performed in 43 patients before open retropubic radical prostatectomy.
  Other Names: Urethral pressure profile measurement

SUMMARY:
Urinary incontinence (UI) is one of the most common complications of radical prostatectomy (RP). Impaired urethral sphincter function is generally considered to be the most important contributing factor of UI however, the mechanism of onset and recovery of urinary continence has not been fully elucidated. In this research, the urodynamic method of Urethral Pressure Profile (UPP) was used to evaluate Functional Urethral Length (FUL) and Maximal Urethral Closure Pressure (MUCP) and correlate with the postprostatectomy continence recovery. Objective of this research is to evaluate preoperative FUL and MUCP as an early continence recovery predictors after open retropubic RP (ORRP).

The research was conducted at the Department of Urology of the University Hospital Centre Zagreb on a group of 43 patients in the period from July 15th , 2019 to May 07th , 2021.The severity of UI and bothersome were assessed using fully validated International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF) and number of pads used in 24h. Patients were interviewed about the use of urinary pads and asked to fill out the ICIQ-UI SF before and 2, 8, 16 and 24 weeks after RP.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with localized prostate cancer
2. Open Retropubic Radical Prostatectomy (ORRP) is planned as a treatment

Exclusion Criteria:

1. Incontinent patients prior to ORRP
2. Previous surgery in the area of the prostatic urethra
3. Previous procedures that can damage the innervation of the pelvis
4. Radiotherapy performed in the pelvic area prior to ORRP
5. Adjuvant radiotherapy in the first postoperative year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients enrolled in the study have prostate cancer.
Enrollment: 43 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Functional Urethral Length as a predictor of Urinary Incontinence | 24 weeks
  Functional Urethral Length (FUL) is measured using Urethral Presssure Profilometry and expressed in mm. The severity of urinary incontinence and bothersome were assessed using fully validated International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF) and number of pads used in 24h. Patients were interviewed about the use of urinary pads and asked to fill out the ICIQ-UI SF before and 2, 8, 16 and 24 weeks after radical prostatectomy. ICIQ-UI SF score ranges: min 0, max 21 (higher score indicating greater severity of symptoms). Cut-off for positive UI, in this research, was 6. Cut-off for positive UI by number of pads used per day was 2.
Maximum Urethral Closure Pressure as a predictor of Urinary Incontinence | 24 weeks
  Maximum Urethral Closure Pressure (MUCP) is measured using Urethral Presssure Profilometry and expressed cmH2O. The severity of urinary incontinence and bothersome were assessed using fully validated International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF) and number of pads used in 24h. Patients were interviewed about the use of urinary pads and asked to fill out the ICIQ-UI SF before and 2, 8, 16 and 24 weeks after radical prostatectomy. ICIQ-UI SF score ranges: min 0, max 21 (higher score indicating greater severity of symptoms). Cut-off for positive UI, in this research, was 6. Cut-off for positive UI by number of pads used per day was 2.

CONTACTS AND LOCATIONS:
Overall Officials: Mirko Bakula, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (1):
- UHC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
IPD that underlie results in a publication (Urethral Pressure Profilometry results, ICIQ-UI SF scoring charts and urinary pads usage) will be available upon the request to Principal Investigator

REFERENCES:
- [Derived] Bakula M, Hudolin T, Kolar Mitrovic H, Kastelan Z. Urethral pressure profile before radical prostatectomy as a predictor of early postoperative continence. Neurourol Urodyn. 2022 Aug;41(6):1431-1439. doi: 10.1002/nau.24978. Epub 2022 Jun 7. PMID 35670263